CLINICAL TRIAL: NCT01406483
Title: Platelet Reactivity in Patients on a Thienopyridine and Awaiting Coronary Artery Bypass Grafting
Acronym: Serial CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Serial CABG
Record Dates: First submitted 2011-07-22; First posted 2011-08-01 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2018-06

CONDITIONS: Complication of Coronary Artery Bypass Graft; Peri-operative Hemorrhage or Hematoma; Post Operative Bleeding
Keywords: Platelet reactivity; CABG; Perioperative and in hospital bleeding
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CABG (Other)
  Interventions: Other: Platelet reactivity assessment

INTERVENTIONS:
Other: Platelet reactivity assessment — Platelet reactivity, as measured by the Chrono-log Lumi-Aggregometer, VerifyNow P2Y12 assay, and Vasodilator Stimulated Phosphoprotein (VASP) flow cytometry assay.

SUMMARY:
The primary objective of this exploratory cohort study is to describe levels of platelet reactivity in patients on a thienopyridine awaiting coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
The recent emergence of platelet reactivity testing as a potential option for evaluating the degree of platelet inhibition promises to add another level of understanding to our concept of CABG-related bleeding. There is an emerging literature that links high levels of platelet reactivity with adverse clinical events, primarily in patients on clopidogrel.

For example, studies of the VerifyNow P2Y12 platelet function assay have shown that Platelet Reactivity Units (PRU) > 235-240 in patients on clopidogrel therapy appears to predict cardiovascular events.15,16 There is a paucity of literature, however, on the use of platelet reactivity testing to predict bleeding events and complications. In other words, if excessively high levels of platelet reactivity predict ischemic events, do excessively low levels of platelet reactivity predict bleeding events? This is an especially relevant question, given the emergence of prasugrel as a therapeutic option.

The investigators therefore propose an exploratory cohort study of patients receiving a thienopyridine (clopidogrel or prasugrel) and undergoing CABG, in order to describe levels of platelet reactivity in such patients by using a variety of platelet function tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old from both genders.
2. Taking maintenance thienopyridine therapy within 5 days of surgery OR received a loading dose of thienopyridine therapy within 48 hours of surgery for CABG.
3. Referred for CABG (which is scheduled to be performed during the current admission).

Exclusion Criteria:

1. Known allergies to aspirin, clopidogrel, or prasugrel.
2. Use of a glycoprotein (GP) IIb/IIIa inhibitor within 8 hours of initial platelet reactivity testing.
3. Patient known to be pregnant or lactating.
4. Patient with known history of bleeding diathesis or currently active bleeding.
5. Platelet count <100,000/mm the day of initial blood draw.
6. Hematocrit <25% the day of initial blood draw.
7. On warfarin therapy at the time of initial blood draw.
8. Known blood transfusion within the preceding 10 days of the blood draw.
9. Patients treated with non-steroidal anti-inflammatory drugs (NSAIDS) within the previous 5 days.
10. Plan for patient to be discharged before undergoing CABG.
11. Any significant medical condition that, in the investigator's opinion, may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Serial levels of platelet reactivity, as assessed with the Chrono-log Lumi-Aggregometer | Duration of hospital stay; average hospital stay of 1 week
  Serial levels of platelet reactivity, as assessed with the Chrono-log Lumi-Aggregometer, which measures levels of light transmittance after stimulation with ADP to estimate levels of platelet aggregation
Perioperative rates of bleeding complications | Duration of hospital stay; average hospital stay of 1 week
  Perioperative rates of bleeding complications:
  1. need for reoperation because of bleeding
  2. need for perioperative red blood cell transfusion (units of packed red blood cells)
  3. rates of TIMI, GUSTO, and nuisance bleeding
  4. quantity of postoperative drainage (mL)

SECONDARY OUTCOMES:
Serial levels of platelet reactivity, as assessed with the VerifyNow P2Y12 assay | Duration of hospital stay; average hospital stay of 1 week
  Serial levels of platelet reactivity, as assessed with the VerifyNow P2Y12 assay, which measures platelet reactivity units (PRUs)
Serial levels of platelet reactivity, as assessed with the Vasodilator Stimulated Phosphoprotein (VASP) assay | Duration of hospital stay; average hospital stay of 1 week
  Serial levels of platelet reactivity, as assessed with the Vasodilator Stimulated Phosphoprotein (VASP) assay, which measures percentage of platelet reactivity inhibition (PRI) by flow cytometry of the VASP-P protein